CLINICAL TRIAL: NCT00316290
Title: Integrated Treatment for Depressed Mothers of ADHD Children
Brief Title: Integrated Parent Training for Treating Depression in Mothers of Children With Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Andrea Chronis-Tuscano, Associate Professor - Psychology, University of Maryland, College Park
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R34MH073567 (NIH); R34MH073567 (NIH); DSIR 84-CTS
Record Dates: First submitted 2006-04-18; First posted 2006-04-20 (Estimated); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Depression; Attention Deficit Disorder With Hyperactivity
Keywords: ADHD; Cognitive Behavioral Therapy; Parent Training
MeSH Terms: conditions — Depression; Attention Deficit Disorder with Hyperactivity

ARMS (2):
- 1 (Experimental): Participants will receive integrated parent training.
  Interventions: Behavioral: Integrated Parent Training
- 2 (Active Comparator): Parents will receive behavioral parent training.
  Interventions: Behavioral: Behavioral Parent Training

INTERVENTIONS:
Behavioral: Integrated Parent Training — Treatment will include behavioral parent training, a course on coping with depression, and cognitive-behavioral therapy targeted at coping with stressful parenting situations. Treatment will include weekly 2-hour sessions for 14 weeks.
  Arms: 1
Behavioral: Behavioral Parent Training — Parents will receive behavioral training. Treatment will include weekly 2-hour sessions for 14 weeks.
  Arms: 2

SUMMARY:
This study will determine the effectiveness of integrated parent training versus standard behavioral parent training in treating depression and stress in mothers of children with attention deficit hyperactivity disorder (ADHD).

DETAILED DESCRIPTION:
ADHD is one of the most common childhood mental disorders. Children with ADHD have impaired functioning in multiple settings, including home and school, and in relationships with peers. Parenting a child with ADHD can be discouraging and stressful. Research has shown that parent-child interactions are more negative among families with ADHD children. Additionally, families with children with ADHD experience increased parental stress, maternal depression, and marital distress, as compared to families with healthy children. These interactions may exacerbate the child's ADHD symptoms. Behavioral parent training has been used to improve parent-child relationships. This study will determine the effectiveness of integrated parent training versus standard behavioral parent training in treating depression and stress in mothers of children with ADHD.

Individuals interested in participating in this open-label study will first undergo an assessment of their eligibility for inclusion in the study. This session will last between 3 and 4 hours and will involve both the mother and the child. If eligible, mothers will be randomly assigned to receive either standard behavioral parent training or an integrated treatment, involving both behavioral parent training and cognitive-behavioral therapy targeted at coping with stressful parenting situations. The integrated treatment will also include a course on coping with depression. Both groups will meet for 2 hours every Wednesday evening for 14 weeks. Childcare will be provided, as well as free treatment for childrens' ADHD symptoms and mothers' depression. Both the child's and the mother's psychological functioning will be assessed upon study completion and at the 3-month follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

Mothers:

* Scores at least 10 on the Beck Depression Inventory (BDI)-II scale on two occasions approximately 1 week apart
* Does not meet criteria for current substance abuse, psychosis, or bipolar disorder, which would likely warrant other immediate treatment

Children:

* Meets DSM-IV criteria for ADHD according to parent and teacher reports on rating scales and parent diagnostic interviews
* Estimated IQ of at least 70
* Aged between 6 and 12 years
* Lives with mother

Exclusion Criteria:

* Child has current Pervasive Development Disorder
* Mothers and children participating in psychosocial treatment that cannot be suspended

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2006-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Maternal depression | Measured post-treatment and at 3-month follow-up

SECONDARY OUTCOMES:
Maternal stress and cognitions | Measured post-treatment and at 3-month follow-up
Child behavior and impairment | Measured post-treatment and at 3-month follow-up
Self-report and observed parenting behaviors | Measured post-treatment and at 3-month follow-up
Family functioning | Measured post-treatment and at 3-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Andrea M. Chronis, PhD, Principal Investigator — University of Maryland, College Park
Locations (1):
- University of Maryland, College Park, College Park, Maryland, United States